CLINICAL TRIAL: NCT04606498
Title: Blood Purification With Seraph® 100 Microbind® Affinity Blood Filter for the Treatment of Severe COVID-19: An Observational Study (PURIFY-OBS-1)
Brief Title: Blood Purification With Seraph 100 Microbind Affinity Blood Filter for Treatment of Severe COVID19 Observational Study
Acronym: PURIFY-OBS-1
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: PURIFY-OBS-1
Record Dates: First submitted 2020-10-26; First posted 2020-10-28 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Covid19
Keywords: Covid19; ICU; Seraph®-100 Microbind® Affinity Blood Filter
MeSH Terms: conditions — COVID-19 | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Biospecimen (blood, urine, sputum, swabs) will be collected at D0, before initiation of extracorporeal treatment, and on study days 1, 2, 3, 4, 7, 28, and 90-180. Since a goal of this study is to recruit as many subjects as possible (predominantly for safety purposes), if a patient is started on Seraph® 100 prior to being recruited for the study, lab collection will begin at the next time point. For example, if a patient is started on Seraph® 100 on a Sunday and the patient is not enrolled until Monday, study day 0 labs will be marked as missing and lab collection will begin on study day 1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1- Retrospective: Retrospective Seraph® 100 - this group will be composed of subjects that were treated with Seraph® 100 after the date of the EUA approval (17 April 2020), but before the date that the study is approved at the study site. A waiver of informed consent will be requested from the Institutional Review Board (IRB) to allow the collection of these retrospective data
  Interventions: Other: Observational
- 2 - Prospective: Prospective Seraph® 100 - To identify prospective Seraph® 100 patients, the individual site investigators will review currently admitted ICU patients for inclusion criteria and exclusion criteria. The study team will then ask the physician caring for the patient to contact the study team should the patient require therapy with Seraph® 100. Additionally, the study team will review the medical records of admitted patients to see if they have recently been started on Seraph. Patients found to meet eligibility will be offered the opportunity to consent and participate in the study. Note that patients that were started on Seraph® 100 before the date of approval but are still admitted, will not be eligible to give biospecimens.
  Interventions: Other: Observational
- 3 - Historical Control: The historical control group will be a sample of convenience, composed of patients admitted to the ICU at participating sites with severe COVID-19 infection, meeting the EUA treatment criteria, but not treated with Seraph® 100 up to the time the PURIFY-OBS protocol is approved at the site. A waiver of informed consent will be requested from the IRB to allow the collection of these retrospective data
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational study only - no intervention

SUMMARY:
This is a multi-center, observational study that will enroll 1) patients with severe COVID-19 who have agreed to undergo therapy with Seraph® 100 under the existing EUA; 2) patients (medical record data) that have been previously treated with the Seraph® 100 after the date of the EUA approval (17 April 2020), but before the date that the study is approved at the study site, and 3) a convenience sample of patients (medical record data) in a historical control group who were admitted to the ICU at participating sites with severe COVID-19 infection, meeting the EUA treatment criteria, but not treated with Seraph® 100 up to the time the PURIFY-OBS protocol is approved at the site

DETAILED DESCRIPTION:
This is a multi-center, observational study that will enroll 1) patients with severe COVID-19 who have agreed to undergo therapy with Seraph® 100 under the existing EUA; 2) patients (medical record data) that have been previously treated with the Seraph® 100 after the date of the EUA approval (17 April 2020), but before the date that the study is approved at the study site, and 3) a convenience sample of patients (medical record data) in a historical control group who were admitted to the ICU at participating sites with severe COVID-19 infection, meeting the EUA treatment criteria, but not treated with Seraph® 100 up to the time the PURIFY-OBS protocol is approved at the site

At the time of protocol approval, data from all patients who have been treated up until that date will be collected retrospectively. Patients who meet the treatment criteria and are identified as candidates for Seraph® 100 with plans for treatment initiation will be enrolled prospectively after informed consent has been obtained. Biospecimen collection (blood, urine, sputum, swabs) will be planned for prospectively enrolled patients at various time-points. However, if subjects do not want to contribute samples, they will be given the option of contributing only their clinical data for analysis. Specific Seraph® 100 treatment procedures will be determined by each individual site. Recommendations for treatment related procedures are provided by the company. Additionally, among sites participating in PURIFY-OBS, all patients who met EUA treatment criteria but were NOT initiated on therapy will be enrolled retrospectively into a historical control group. Procedures for identifying study subjects will be as follows:

Retrospective Seraph® 100 As noted in the inclusion/exclusion criteria, this group will be composed of subjects that were treated with Seraph® 100 after the date of the EUA approval (17 April 2020), but before the date that the study is approved at the study site. To identify patients, the site investigator will query 1) institution's electronic medical record for critical ill patients treated with Seraph® 100 and 2) attending intensive care physicians and nephrologists who have provided care to critically ill patients with COVID-19. A waiver of informed consent will be requested from the Institutional Review Board (IRB) to allow the collection of these retrospective data.

Prospective Seraph® 100 To identify prospective Seraph® 100 patients, the individual site investigators will review currently admitted ICU patients for inclusion criteria #1and #2 (see above). The study team will then ask the physician caring for the patient to contact the study team should the patient require therapy with Seraph® 100. Additionally, the study team will review the medical records of admitted patients to see if they have recently been started on Seraph. Patients found to meet inclusion/exclusion criteria (or their LARs) will be offered the opportunity to sign an informed consent and participate in the study. Note that patients that were started on Seraph® 100 before the date of approval for a study site, but are still admitted, will not be eligible to give biospecimens. However, they will be given the option of signing an informed consent so that their data can be used in the study.

Historical Control Our historical control group will be a sample of convenience, composed of patients admitted to the ICU at participating sites with severe COVID-19 infection, meeting the EUA treatment criteria, but not treated with Seraph® 100 up to the time the PURIFY-OBS protocol is approved at the site. The individual site investigators will be responsible for querying their institution's electronic medical records to identify critically ill patients with COVID-19 admitted from the date of EUA approval (17 April 2020) until the date the protocol was approved at their study site. These records will then be further examined by the local study team to ensure that the patients meet the inclusion/exclusion criteria detailed above. Note that patients will be excluded if they are still admitted to the hospital on or after the date that the protocol was approved at that study site. A waiver of informed consent will be requested from the Institutional Review Board (IRB) to allow the collection of these retrospective data.

Study Timeline Each included subject's medical record will be reviewed from the time of hospital admission through hospital discharge. Enrollment will be conducted over a 2-year period (up to 200 patients total including both retrospective and prospective patients). For prospective patients who consent, biospecimen (blood, urine, sputum) will be collected before initiation of extracorporeal treatment, 1 hour following treatment, as well as days 1, 2, 3, 4, 7, 28 and 90-180

ELIGIBILITY:
Inclusion Criteria:

Prospective Seraph® 100

1. Subject must be 18 years of age
2. Per the FDA Approve EUA:

Subject must have confirmed COVID-19 infection and be admitted to the ICU with confirmed or imminent respiratory failure and any one of the following conditions:

1. Early acute lung injury (ALI)/early acute respiratory distress syndrome (ARDS); or
2. Severe disease, defined as:

   1. Dyspnea,
   2. Respiratory frequency ≥ 30/min,
   3. Blood oxygen saturation ≤ 93%,
   4. Partial pressure of arterial oxygen to fraction of inspired oxygen ratio <300, and/or
   5. Lung infiltrates > 50% within 24 to 48 hours; or
3. Life-threatening disease, defined as:

   1. Respiratory failure,
   2. Septic shock, and/or
   3. Multiple organ dysfunction or failure. 2. Prospective study patients (or their Legally Authorized Representative (LAR)) provides informed consent. Patients or their legally authorized representative will be consented in their main language if they are not fluent in English.

   3. Prospective study patient is willing to complete all study visits as required by the protocol 4. For Military Treatment Facility (MTF) enrollment only - must be DEERS eligible for care at the MTF

Retrospective Seraph® 100

1. Subject must be 18 years of age
2. Per the FDA Approve EUA:

   Subject must have confirmed COVID-19 infection and be admitted to the ICU with confirmed or imminent respiratory failure and any one of the following conditions:
   1. Early acute lung injury (ALI)/early acute respiratory distress syndrome (ARDS); or
   2. Severe disease, defined as:

      1. Dyspnea,
      2. Respiratory frequency ≥ 30/min,
      3. Blood oxygen saturation ≤ 93%,
      4. Partial pressure of arterial oxygen to fraction of inspired oxygen ratio <300, and/or
      5. Lung infiltrates > 50% within 24 to 48 hours; or
   3. Life-threatening disease, defined as:

      1. Respiratory failure,
      2. Septic shock, and/or
      3. Multiple organ dysfunction or failure.
3. Treated with Seraph® 100 from 17 April 2020 (date of EUA approval) to the date of study approval at the study site.

Historical Control

1. Subject must be 18 years of age
2. Per the FDA Approve EUA:

   Subject must have confirmed COVID-19 infection and be admitted to the ICU with confirmed or imminent respiratory failure and any one of the following conditions:
   1. Early acute lung injury (ALI)/early acute respiratory distress syndrome (ARDS); or
   2. Severe disease, defined as:

      1. Dyspnea
      2. Respiratory frequency ≥ 30/min,
      3. Blood oxygen saturation ≤ 93%,
      4. Partial pressure of arterial oxygen to fraction of inspired oxygen ratio <300, and/or
      5. Lung infiltrates > 50% within 24 to 48 hours; or
   3. Life-threatening disease, defined as:

   <!-- -->

   1. Respiratory failure,
   2. Septic shock, and/or
   3. Multiple organ dysfunction or failure.
3. Hospitalized from 20 January 2020 to the date of study approval at the study site.

Exclusion Criteria:

Prospective

1. Unwilling to provide informed consent
2. Unable to provide informed consent and no LAR available to provide permission

Retrospective No specific exclusion criteria. However, patients treated with Seraph® 100 prior to approval of the study at a site and who remains admitted to the hospital at the time the study is approved, will be given the opportunity to participate in the study by signing consent for their health data to be collected (and not biospecimens).

Historical Controls:

Patients who remain admitted to the hospital at the time that the study is approved at the study site will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This multi-center, observational study will attempt to recruit all patients treated with the Seraph® 100 under EUA #200165 in the United States at both civilian and military hospitals.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Time spent on medications used to increase blood pressure | Measure from start of medication (day 0) to day 28 of study
  list type of medication and length of medication for Blood pressure

SECONDARY OUTCOMES:
Time spent on mechanical ventilation | From intubation date through extubation or day 28 of study
  Length of time on ventilator
Time spent in the intensive care unit (ICU) | admission to ICU (day 0) through ICU discharge or up to day 28 of study
  Length of time patient in the ICU
Time spent in the hospital | from hospital admission (day 0) to discharge or up to day 28
  Length of time patient was hospitalized
Time spent on dialysis | Start of dialysis treatment (day 0) to end of dialysis or up to day 28
  length of time patient required dialysis
Mortality | From diagnosis of Covid (day 0) to date of death up to day 28
  survival

CONTACTS AND LOCATIONS:
Overall Officials: Ian Stewart, MD, Principal Investigator — USUHS/WRNMMC
Locations (14):
- United States (14):
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - University of Colorado Hospital, Aurora, Colorado
  - Advent Health, Orlando, Florida
  - Southeast Georgia Health System - Brunswick Campus, Brunswick, Georgia
  - Eisenhower Army Medical Center (EAMC), Fort Gordon, Georgia
  - Ian Stewart, Bethesda, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Forrest General Hospital, Hattiesburg, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baylor Scott & White, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Methodist Hospital, San Antonio, Texas
  - University Of Texas Health San Antonio (UTHSA)- University Health, San Antonio, Texas
  - Brooke Army Medical Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided